CLINICAL TRIAL: NCT05745896
Title: A Telemedicine Prenatal Care Model on Low Risk Pregnants: An Effectiveness Randomized Clinical Trial (The m@Mae-e Study)
Brief Title: A Telemedicine Prenatal Care Model on Low Risk Pregnants: The m@Mae-e Study
Acronym: m@mae-e
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Talita Colombo (Other)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other); McMaster University (Other); VU University of Amsterdam (Other); Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor-Investigator, Talita Colombo, Talita Colombo, MD, MSc - Principal Investigator, Federal University of Health Science of Porto Alegre
Organization: Federal University of Health Science of Porto Alegre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 48740621.9.0000.5335
Record Dates: First submitted 2022-07-31; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Pregnancy; Mental Disorders; COVID-19 Pandemic; Prenatal Stress
Keywords: prenatal care; covid-19; telemedicine; low risk prenatal line of care; health policy; randomized clinical trial
MeSH Terms: conditions — Mental Disorders; COVID-19

STUDY DESIGN:
Intervention Model Description: A superiority randomized clinical trial (RCT), comparing usual care against telemedicine prenatal care. The allocation ratio is a proportion of 1:1 and the maximum follow-up will last 41 weeks (6 weeks pregnancy to 6 week postpartum).
Who Masked: Outcomes Assessor
Masking Description: Adequate masking will be tentatively done by ensuring the allocation concealment, mitigating possibilities of masking violations by outcomes assessors. In addition, an electronic case report form system will be used in a de-identified manner. Only study's chairs will have access to codes. Finally, interim and final analysis will be done in the same manner after dataset locking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Pregnants at usual care attending appointments in-person.
  Interventions: Other: Face-to-face appointment
- Telemedicine Prenatal Care (Experimental): Pregnants under telemedicine based group attending at least 6 in-person outpatient clinic appointments and the remaining ones (i.e., 3) online.
  Interventions: Other: Telemedicine appointment; Other: Face-to-face appointment

INTERVENTIONS:
Other: Telemedicine appointment — Three online appointments for pregnancy monitoring at prenatal care.
  Arms: Telemedicine Prenatal Care
Other: Face-to-face appointment — Six to nine face-to-face appointments for pregnancy monitoring at prenatal care.

SUMMARY:
This study will compare the effectiveness of a prenatal care supported by telemedicine against usual care in low-risk pregnant women. The investigators will follow-up women in a gestational age of 6 weeks up to 41 weeks, and 6 postpartum weeks. The primary outcome is the anxiety level estimated by the General Anxiety Scale 7 scale (GAD-7 Scale).

DETAILED DESCRIPTION:
This is a pragmatic, effectiveness, superiority randomized clinical trial (RCT), in which low risk pregnants will be randomized to a prenatal care program supported by telemedicine or usual care in an allocation ratio of 1:1. The follow-up period will last 41 weeks from inception (i.e., 6 to 13 weeks of gestational age) to pregnancy and a extension period of 6 weeks in the postpartum stage. The investigators settled anxiety levels estimated by the General Anxiety Scale 7 scale as primary outcome in a between-groups mean difference after the 3rd trimester. Secondary outcomes include: delivery mode, obstetric events and fetal and neonatal variables of epidemiological surveillance interest (birth weight, birth height and APGAR score; maternal, fetal and neonatal fatal and non-fatal events). The interventions will occur as follows: for usual care, all appointments (at least 9 outpatient clinic visits) will be carried forward in person by a senior obstetrician. Patients randomized for the telemedicine supported group should will attend at least 6 in person and 3 online appointments. All pregnant women will receive the standardized care throughout the study. The sample size calculation was based on the primary outcome, assuming between-groups mean difference of 4 points plus a 4-points standard deviation, at a statistical of 80% and a two-tailed 5% type I error. Further, a 15% of addition was done for potential impairments during the follow-up, ending in 30 patients per group. The m@mae-e study's setting will be the at Santa Casa de Misericórdia, (Porto Alegre, Brazil).

ELIGIBILITY:
Inclusion Criteria:

* Low-risk pregnant (as classified an attending physician and/or the study's obstetrician);
* Gestational age less at 13 weeks or more in the moment of the first appointment;
* Portuguese native speaker.

Exclusion Criteria:

* Pregnant involving: hypertension or diabetes mellitus (any type) previous diagnosis;
* Obesity (BMI equal or greater than 35 m/kg2;
* Previous diagnosis of severe Sars-CoV-2 2019-related (COVID-19) infection which needed hospitalization;
* Previous thromboembolic event;
* Acute or chronic hematological events/diseases; use of anticoagulants or anti platelet aggregation drugs;
* Chronic cardiovascular, lung or kidney disease and cancer requiring treatment;
* Immunosuppression state;
* Severe mental disorder - major depression, generalized anxiety (and others anxiety-related disorders), bipolar disorder, schizophrenia and personality-related disorders in an uncontrolled manner for at least 1 year;
* At least more than one abortion;
* History of premature birth;
* An enrolled patient living in the same house;
* Plan to move the city.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety levels in usual care and telemedicine support care groups from inception until the final of the prenatal care (6 weeks postpartum). | First measure at baseline, last measure at birth time
  Mean between-group differences in General Anxiety Disorder (GAD-7) scale scores.
Anxiety levels in usual care and telemedicine support care groups from inception until the final of the postpartum period (6 weeks postpartum). | First measure at baseline, last measure at the end of postpartum period (6 week postpartum).
  Mean between-group differences in General Anxiety Disorder (GAD-7) scale scores.

SECONDARY OUTCOMES:
Secondary analysis of anxiety levels between usual care and telemedicine support care groups. | Repeated, full comparisons estimates at baseline; 10-12th weeks of pregnancy; 18-24 weeks of pregnancy and 34-36 weeks of pregnancy as well as the postpartum period (4-6 week postpartum)
  Mean between-groups differences in General Anxiety Disorder (GAD-7) scale scores.
Maternal fatal and non-fatal outcomes | Assesed at birth
  Cumulative incidence of gestational diabetes diagnosis; high blood pressure events (pre-eclampsia and eclampsia); severe anemia; need to forward to high-risk prenatal care program; cardiovascular events with or without hospitalization; cardiovascular attributable death during pregnancy and postpartum period; maternal attributable underlying cause of death; all-cause mortality.
Fetal and neonatal fatal and non-fatal outcomes | Assesed at birth
  Cumulative incidence and mean difference between-groups of: gestational age at birth; birth weight; APGAR score; neonatal intensive care unit (ICU) admission; death by intentional and unintentional abortion; events related to underlying causes of fetal and neonatal periods; fatal events related to underlying causes of fetal and neonatal events
Quality of life levels between usual care and telemedicine support care | Repeated, full comparisons estimates at baseline; 10-12th weeks of pregnancy; 18-24 weeks of pregnancy and 34-36 weeks of pregnancy as well as the postpartum period (4-6 week postpartum)
  Mean between-groups differences in the Portuguese validated EuroQoL 5D scores (EQ-5D).

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Helal, MSc, PhD, Study Chair — Federal University of Rio Grande do Sul; Airton T Stein, MD, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Irmandade da Santa Casa de Misericórdia de Porto Alegre (ISCMPA), Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We added an individual participant data sharing policy (IPD data-sharing) and tabular results will be displayed in this CT.gov in a 12-month range after our primary completion (PC) at max. Third parties interested to use the m@mae-e data should contact the study chair and the study's PI. IPD will be released in a public and safe repository in a de identified manner. Altogether to the raw data, individuals will have access to case report files, the study protocol, materials, SAP and codes.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after primary completion date, for at least 10 years.
Access Criteria: Open access accompanied by a disclosure form of potential conflicts of interest and Term of Agreement to not make misuse of the data.
URL: https://osf.io/6xzyf/

REFERENCES:
- [Background] Colombo T, Todeschini LB, Orlandini M, Nascimento HD, Gabriel FC, Alves RJV, Stein AT. Low-Risk Antenatal Care Enhanced by Telemedicine: A Practical Guideline Model. Rev Bras Ginecol Obstet. 2022 Sep;44(9):845-853. doi: 10.1055/s-0042-1753505. Epub 2022 Jul 19. PMID 35853473
- [Background] Stein C, Helal L, Migliavaca CB, Sangalli CN, Colpani V, Raupp da Rosa P, Beck-da-Silva L, Rohde LE, Polanczyk CA, Falavigna M. Are the recommendation of sodium and fluid restriction in heart failure patients changing over the past years? A systematic review and meta-analysis. Clin Nutr ESPEN. 2022 Jun;49:129-137. doi: 10.1016/j.clnesp.2022.03.032. Epub 2022 Apr 6. PMID 35623804
- See also: Repository for study's management. — https://osf.io/6xzyf/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT05745896/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT05745896/ICF_001.pdf